CLINICAL TRIAL: NCT00459121
Title: Assessment of Feasibility and Safety of the Addition of ZD6474 (Zactima) to Carboplatin and Paclitaxel Administered Neo-Adjuvantly in Stage IB, II and T3, N1 Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Vandetanib, Carboplatin, and Paclitaxel in Treating Patients With Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shirish M. Gadgeel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000539273; P30CA022453 (NIH); WSU-2006-122 (Other: Barbara Ann Karmanos Cancer Institute); WSU-011807MP2F (Other: Wayne State University - Human Investigation Committee); WSU-0612004427 (Other: Wayne State University - Human Investigation Committee); ZENECA-IRUSZACT0029
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2012-12-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; vandetanib; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zactima, Paclitaxel, Carboplatin (Experimental): Zactima- 100 mg orally daily, starting on day 1 of cycle 1. Paclitaxel- 200mg/m2 IV, every 3 weeks starting on day 1 of cycle 1. Carboplatin AUC6 IV, every 3 weeks starting on day 1 of cycle 1 Duration of each cycle: 21 days. The last dose of zactima will be on the first day of the last cycle.
  Neoadjuvant Surgery: Surgical resection of the tumor will be performed after the resolution of all the adverse effects from the last cycle of treatment but no earlier than 3 weeks after the last cycle of treatment.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: Zactima; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: carboplatin — Carboplatin AUC6 IV, every 3 weeks starting on day 1 of cycle 1
  Other Names: Paraplatin ®
Drug: paclitaxel — Paclitaxel- 200mg/m2 IV, every 3 weeks starting on day 1 of cycle 1.
  Other Names: Taxol ®; Onxal TM
Drug: Zactima — Zactima- 100 mg orally daily, starting on day 1 of cycle 1.
  Other Names: Caprelsa; ZD6474; Vandetanib
Procedure: neoadjuvant therapy — Neoadjuvant surgery: Surgical resection of the tumor will be performed after the resolution of all the adverse effects from the last cycle of treatment but no earlier than 3 weeks after the last cycle of treatment.
  Other Names: R0 Resection

SUMMARY:
RATIONALE: Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vandetanib together with chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving vandetanib together with carboplatin and paclitaxel works in treating patients with stage I, stage II, or stage III non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of neoadjuvant vandetanib in combination with carboplatin and paclitaxel in patients with resectable stage IB, II, or IIIA non-small cell lung cancer.

Secondary

* Assess the 30-day postoperative mortality rate in these patients.
* Assess the toxicity of this regimen in these patients.
* Determine the percentage of patients who complete all planned courses of therapy.
* Assess the clinical response rate in patients treated with this regimen.
* Assess the pathologic complete response rate in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral vandetanib once daily on days 1-21. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 3 courses.

Patients undergo surgery at least 3 weeks after the last course of chemotherapy.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), meeting 1 of the following staging criteria:

  * Stage IB or II disease
  * T3, N0-1 disease (stage IIIA)
* Deemed a surgical candidate
* No prior lung cancer (NSCLC or small cell lung cancer)

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of severe or uncontrolled systemic disease or any concurrent condition that, in the opinion of the investigator, would preclude study compliance
* No peripheral neuropathy ≥ grade 2
* No hemoptysis within the past 12 weeks
* No spontaneous bleeding within the past 12 weeks
* No clinically significant cardiac event (e.g., NYHA class II-IV heart disease, myocardial infarction) within the past 3 months
* No history of asymptomatic sustained ventricular tachycardia or arrhythmia that is symptomatic or requires treatment, including any of the following:

  * Multifocal premature ventricular contractions
  * Bigeminy
  * Trigeminy
  * Ventricular tachycardia
  * Uncontrolled atrial fibrillation

    * Atrial fibrillation controlled with medication allowed
* No history of QTc prolongation as a result from other medication that required discontinuation of that medication
* No congenital long QT syndrome or first-degree family relative with an unexplained death before the age of 40
* No left bundle branch block
* No QTc with Bazett's correction that is unmeasurable or QTc ≥ 480 milliseconds on screening ECG

  * Patients with QTc ≥ 480 milliseconds on screening ECG may have ECG repeated twice

    * Average QTc from the 3 screening ECG's must be < 480 milliseconds
* No uncontrolled hypertension (systolic BP > 160 mm Hg or diastolic BP > 100 mm Hg)
* No active diarrhea or active gastrointestinal disease that may affect the absorption of study drugs or ability to tolerate study drugs
* No other malignancy within the past 3 years except in situ cervical carcinoma or adequately treated basal cell or squamous cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since major surgery and recovered
* No prior carboplatin, paclitaxel, or vandetanib
* More than 30 days since prior investigational agents
* More than 2 weeks since prior and no concurrent drugs that induce CYP3A4 including, but not limited to, any of the following:

  * Rifampin
  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
* No medication that may cause QTc prolongation or induce torsades de pointes for 2 weeks prior to beginning study treatment, during, and for 2 weeks after completion of study treatment
* No concurrent combination antiretroviral treatment for HIV-positive patients
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unable to enroll patients in a timely fashion. The decision was made to close the study after consulting with AstraZeneca.
Pre-assignment Details: Feasibility and safety.
Period: Overall Study
Arm/Group | Zactima, Paclitaxel, Carboplatin
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zactima, Paclitaxel, Carboplatin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Resection (R0) Rate
Time Frame: Following three cycles of pre-operative zactima and carboplatin/paclitaxel
Population: No analysis was completed only 2 patients enrolled, study closed due to slow accrual.
Groups:
- Zactima+Carboplatin & Paclitaxel-assess Feasibility & Safety: Study closed before an evaluable number of participants could be accrued. No summary of statistics will be collected for two participants, per the statistician.
Arm/Group | Zactima+Carboplatin & Paclitaxel-assess Feasibility & Safety
Number analyzed (Participants) | 0

2. Secondary Outcome: Post-Operative Mortality Rate
Time Frame: at 30 days
Population: No analysis was completed only 2 patients enrolled, study closed due to slow accrual.
Arm/Group | Zactima, Paclitaxel, Carboplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess Toxicity of This Regimen and the Percentage of Patients Completing All Planned Cycles of Therapy
Description: Serum chemistry includes Albumin, alkaline phosphatase, total bilirubin, bicarbonate, BUN, calcium, chloride, creatinine, glucose, potassium, total protein, SGOT [AST], SGPT [ALT], sodium, laboratory tests should be done on a weekly basis for the first cycle. After the first cycle laboratory tests should be done within 72 hours of each dose of carboplatin/paclitaxel.
Time Frame: Weekly for the first cycle; Thereafter within 72 hours of each dose of carboplatin/paclitaxel
Population: No analysis was completed only 2 patients enrolled, study closed due to slow accrual.
Arm/Group | Zactima, Paclitaxel, Carboplatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Assess the Clinical Response Rate of the Proposed Pre-operative Regimen
Description: Patients will undergo tumor evaluation when all of the three cycles have been completed unless the treating physician has concerns regarding tumor progression. If the patient has undergone tumor evaluation prior to the last cycle the patient will require repeat tumor assessment within 4 weeks of completion of the last cycle of therapy
Time Frame: End of three cycles of treatment
Population: No analysis was completed only 2 patients enrolled, study closed due to slow accrual.
Arm/Group | Zactima, Paclitaxel, Carboplatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Assess the Complete Pathologic Complete Response (CR) Rate With This Regimen.
Description: Evaluation of the number of patients who have no evidence of tumor in the resected tumor.
Time Frame: 30 days post surgery
Population: No analysis was completed only 2 patients enrolled, study closed due to slow accrual.
Arm/Group | Zactima, Paclitaxel, Carboplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Zactima+Carboplatin & Paclitaxel-assess Feasibility & Safety
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zactima+Carboplatin & Paclitaxel-assess Feasibility & Safety (N=2)
Decreased ANC (Blood and lymphatic system disorders) | 2 (2)
Cough (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Bicarbonate (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased WBC count (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Decreased hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a single center study. We did not accrue enough particpants in a timely fashion and a joint decision was made with AstraZeneca to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No